CLINICAL TRIAL: NCT01225562
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Group, Multinational Trial, to Assess the Prevention of Thrombotic Events With Ticagrelor Compared to Placebo on a Background of Acetyl Salicylic Acid (ASA) Therapy in Patients With History of Myocardial Infarction
Brief Title: Prevention of Cardiovascular Events (eg, Death From Heart or Vascular Disease, Heart Attack, or Stroke) in Patients With Prior Heart Attack Using Ticagrelor Compared to Placebo on a Background of Aspirin
Acronym: PEGASUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D5132C00001; 2009-017242-30 (EudraCT Number)
Record Dates: First submitted 2010-07-09; First posted 2010-10-21 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-12

CONDITIONS: Myocardial Infarction; Cardiovascular Death; Atherothrombosis; Stroke
Keywords: Heart attack; Heart Disease; Acute coronary syndrome; ACS; Cardiovascular Disease
MeSH Terms: conditions — Myocardial Infarction; Thrombosis; Stroke; Heart Diseases; Acute Coronary Syndrome; Cardiovascular Diseases | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): Oral Treatment
  Interventions: Drug: Ticagrelor 90 mg
- 2 (Experimental): Oral Treatment
  Interventions: Drug: Ticagrelor 60 mg
- 3 (Placebo Comparator): Oral Treatment
  Interventions: Drug: Ticagrelor Placebo

INTERVENTIONS:
Drug: Ticagrelor 90 mg — Oral dose twice a day
  Arms: 1
Drug: Ticagrelor 60 mg — Oral dose twice a day
  Arms: 2
Drug: Ticagrelor Placebo — Oral dose twice a day
  Arms: 3

SUMMARY:
This study is being carried out to see if a new drug called ticagrelor given twice daily in addition to the ASA therapy decreases the frequency of cardiovascular events (e.g., death from heart disease, heart attack, or stroke).

ELIGIBILITY:
Inclusion Criteria:

* Person who had a heart attack within 1 - 3 years ago and at least one additional risk factor: Age ≥ 65 years old, Diabetes requiring medication, Documented history of 2nd prior MI (>1 year ago). Angiographic evidence of multivessel CAD, and / or Chronic, non-end stage renal dysfunction.
* Females of child-bearing potential must have a negative pregnancy test at enrollment
* Persons who are currently taking aspirin between 75 and 150 mg once daily

Exclusion Criteria:

* Persons who are being treated with agents inhibiting blood clotting if the agent cannot be stopped at study start
* Persons who have planned coronary, cerebrovascular, or peripheral arterial Revascularization (invasive surgery) at study start
* Persons with known bleeding disorders
* Persons who need chronic oral anticoagulant therapy or chronic low-molecular-weight heparin
* Persons with a history of ischemic stroke
* Persons with a history of intracranial bleeding at any time, a tumor or blood vessel abnormality in the brain and/or spinal cord at any time, a history of surgery involving the brain or spinal cord within the last 5 years, or a history of bleeding from the gastrointestinal tract (eg, esophagus, stomach, colon, rectum) within the last 6 months or a major surgery within the last 30 days.
* Persons considered to be at risk of bradycardic events unless already treated with a permanent pacemaker
* Persons who have had open heart surgery within the past 5 years, unless the person had a heart attack after the surgery
* Persons with known severe liver disease
* Persons with kidney failure requiring dialysis
* Persons with life expectancy < 1 year

Ages: 50 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21379 (Actual)
Dates: Start 2010-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Braunwald, MD, Study Chair — The TIMI Study Group; Marc Sabatine, MD, MPh, Principal Investigator — The TIMI Study Group
Locations (827):
- United States (250):
  - Research Site, Alexander City, Alabama
  - Research Site, Athens, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Sheffield, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Jonesboro, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Alhambra, California
  - Research Site, Anaheim, California
  - Research Site, Bakersfield, California
  - Research Site, Fountain Valley, California
  - Research Site, La Mesa, California
  - Research Site, Larkspur, California
  - Research Site, Lomita, California
  - Research Site, Los Angeles, California
  - Research Site, Modesto, California
  - Research Site, Newport Beach, California
  - Research Site, Oakland, California
  - Research Site, Oceanside, California
  - Research Site, San Diego, California
  - Research Site, San Marino, California
  - Research Site, Santa Rosa, California
  - Research Site, Ventura, California
  - Research Site, Westlake Village, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Loveland, Colorado
  - Research Site, Hartford, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boca Raton, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Crystal River, Florida
  - Research Site, Davie, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Largo, Florida
  - Research Site, Leesburg, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Naples, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orlando, Florida
  - Research Site, Pannama City, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Safety Harbor, Florida
  - Research Site, Sarasota, Florida
  - Research Site, South Miami, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, The Villages, Florida
  - Research Site, Wellington, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Cumming, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Boise, Idaho
  - Research Site, Aurora, Illinois
  - Research Site, Bannockburn, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Melrose Park, Illinois
  - Research Site, Normal, Illinois
  - Research Site, Rock Island, Illinois
  - Research Site, Avon, Indiana
  - Research Site, Elkhart, Indiana
  - Research Site, Fort Wayne, Indiana
  - Research Site, Franklin, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Munster, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Hutchinson, Kansas
  - Research Site, Crestview Hills, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Covington, Louisiana
  - Research Site, Minden, Louisiana
  - Research Site, New Iberia, Louisiana
  - Research Site, Opelousas, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Slidell, Louisiana
  - Research Site, Auburn, Maine
  - Research Site, Bangor, Maine
  - Research Site, Biddeford, Maine
  - Research Site, South Portland, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Oxon Hill, Maryland
  - Research Site, Salisbury, Maryland
  - Research Site, Ayer, Massachusetts
  - Research Site, Boston, Massachusetts
  - Research Site, Burlington, Massachusetts
  - Research Site, Haverhill, Massachusetts
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Alpena, Michigan
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Grand Blanc, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Jackson, Michigan
  - Research Site, Lapeer, Michigan
  - Research Site, Marquette, Michigan
  - Research Site, Petoskey, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Saginaw, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Ypsilanti, Michigan
  - Research Site, Baxter, Minnesota
  - Research Site, Duluth, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Robbinsdale, Minnesota
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Biloxi, Mississippi
  - Research Site, Tupelo, Mississippi
  - Research Site, Columbia, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Billings, Montana
  - Research Site, Great Falls, Montana
  - Research Site, Kalispell, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Papillion, Nebraska
  - Research Site, Reno, Nevada
  - Research Site, Bridgewater, New Jersey
  - Research Site, Elizabeth, New Jersey
  - Research Site, Elmer, New Jersey
  - Research Site, Haddon Heights, New Jersey
  - Research Site, Linden, New Jersey
  - Research Site, Mine Hill, New Jersey
  - Research Site, Newark, New Jersey
  - Research Site, Ridgewood, New Jersey
  - Research Site, Somerset, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Buffalo, New York
  - Research Site, Cortlandt Manor, New York
  - Research Site, Mineola, New York
  - Research Site, New Windsor, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Saratoga Springs, New York
  - Research Site, Southampton, New York
  - Research Site, Stony Brook, New York
  - Research Site, The Bronx, New York
  - Research Site, Williamsville, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Burlington, North Carolina
  - Research Site, Cary, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Morganton, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Rocky Mount, North Carolina
  - Research Site, Sanford, North Carolina
  - Research Site, Smithfield, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Grand Forks, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Fairfield, Ohio
  - Research Site, Mansfield, Ohio
  - Research Site, Sandusky, Ohio
  - Research Site, Springfield, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Youngstown, Ohio
  - Research Site, Zanesville, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Bend, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, Beaver, Pennsylvania
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Chambersburg, Pennsylvania
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Johnstown, Pennsylvania
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Langhorne, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Scranton, Pennsylvania
  - Research Site, Sellersville, Pennsylvania
  - Research Site, West Chester, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Florence, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Watertown, South Dakota
  - Research Site, Germantown, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Oak Ridge, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Georgetown, Texas
  - Research Site, Grapevine, Texas
  - Research Site, Houston, Texas
  - Research Site, Katy, Texas
  - Research Site, Kingwood, Texas
  - Research Site, McAllen, Texas
  - Research Site, Plano, Texas
  - Research Site, Round Rock, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tomball, Texas
  - Research Site, Tyler, Texas
  - Research Site, Victoria, Texas
  - Research Site, Provo, Utah
  - Research Site, Burlington, Vermont
  - Research Site, Alexandria, Virginia
  - Research Site, Charlottesville, Virginia
  - Research Site, Danville, Virginia
  - Research Site, Falls Church, Virginia
  - Research Site, Lynchburg, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Winchester, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Everett, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Green Bay, Wisconsin
  - Research Site, Wausau, Wisconsin
- Argentina (21):
  - Research Site, Bahía Blanca
  - Research Site, Buenos Aires
  - Research Site, Ciudad Autonoma de BA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Ciudadela
  - Research Site, Coronel Suárez
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Haedo
  - Research Site, La Plata
  - Research Site, Mar del Plata
  - Research Site, Ramos Mejía
  - Research Site, Rosario
  - Research Site, Rosario Santa Fe
  - Research Site, San Luis
  - Research Site, San Miguel de Tucumán
  - Research Site, San Nicolás
  - Research Site, San Salvador de Jujuy
  - Research Site, Santa Fe
  - Research Site, Santa Fé
  - Research Site, Zárate
- Australia (28):
  - Research Site, Adelaide
  - Research Site, Ashford
  - Research Site, Auchenflower
  - Research Site, Ballarat
  - Research Site, Bruce
  - Research Site, Chermside
  - Research Site, Clayton
  - Research Site, Concord
  - Research Site, East Saint Kilda
  - Research Site, Elizabeth Vale
  - Research Site, Epping
  - Research Site, Fremantle
  - Research Site, Geelong
  - Research Site, Gosford
  - Research Site, Greenslopes
  - Research Site, Herston
  - Research Site, Joondalup
  - Research Site, Kingswood
  - Research Site, Kogorah
  - Research Site, Launceston
  - Research Site, Melbourne
  - Research Site, Nedlands
  - Research Site, New Lambton Heights
  - Research Site, Richmond
  - Research Site, St Leonards
  - Research Site, Wollongong
  - Research Site, Woodville
  - Research Site, Woolloongabba
- Belgium (26):
  - Research Site, Aalst
  - Research Site, Antwerp
  - Research Site, Bonheiden
  - Research Site, Bouge
  - Research Site, Brasschaat
  - Research Site, Brussels
  - Research Site, Brussels (Anderlecht)
  - Research Site, Brussels (Jette)
  - Research Site, Brussels (Woluwé-St-Lambert)
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Huy
  - Research Site, La Louvière
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Mechelen
  - Research Site, Mol
  - Research Site, Ottignies
  - Research Site, Roeselare
  - Research Site, Tienen
  - Research Site, Turnhout
  - Research Site, Yvoir
  - Research Site, Zottegem
- Brazil (20):
  - Research Site, Aracaju
  - Research Site, Belo Horizonte
  - Research Site, Blumenau
  - Research Site, Brasília
  - Research Site, Campina Grande do Sul
  - Research Site, Campinas
  - Research Site, Campo Grande
  - Research Site, Curitiba
  - Research Site, Goiânia
  - Research Site, Maceió
  - Research Site, Marília
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, S.J.Rio Preto
  - Research Site, Salvador
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
  - Research Site, Uberlândia
  - Research Site, Votuporanga
- Bulgaria (11):
  - Research Site, Dimitrovgrad
  - Research Site, Gotse Delchev
  - Research Site, Pernik
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Razlog
  - Research Site, Rousse
  - Research Site, Sevlievo
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
- Canada (45):
  - Research Site, Edmonton, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, New Westminster, British Columbia
  - Research Site, Penticton, British Columbia
  - Research Site, Surrey, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Moncton, New Brunswick
  - Research Site, Saint John, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Cornwall, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Gatineau, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Lévis, Quebec
  - Research Site, Longueuil, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Saint-Georges, Quebec
  - Research Site, Saint-Jérôme, Quebec
  - Research Site, Saint-Lambert, Quebec
  - Research Site, Terrebonne, Quebec
  - Research Site, Thetford-Mines, Quebec
  - Research Site, Val-d'Or, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Chile (7):
  - Research Site, Concepción
  - Research Site, Osorno
  - Research Site, Rancagua
  - Research Site, Santiago
  - Research Site, Santiago Centro
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (13):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Lanzhou
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shengyang
  - Research Site, Shenyang
  - Research Site, Taiyuan
  - Research Site, Wuhan
  - Research Site, Xi'an
- Colombia (10):
  - Research Site, Armenia
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Bogotá D.C.
  - Research Site, Bucaramanga
  - Research Site, Cali
  - Research Site, Cartagena
  - Research Site, Manizales
  - Research Site, Medellín
  - Research Site, Medillin
- Czechia (21):
  - Research Site, Brno
  - Research Site, Chomutov
  - Research Site, Čáslav
  - Research Site, Česká Lípa
  - Research Site, Český Krumlov
  - Research Site, Havířov
  - Research Site, Kroměříž
  - Research Site, Kyjov
  - Research Site, Liberec
  - Research Site, Mariánské Lázně
  - Research Site, Ostrava
  - Research Site, Ostrava-Poruba
  - Research Site, Pelhřimov
  - Research Site, Prague
  - Research Site, Příbram
  - Research Site, Slaný
  - Research Site, Teplice
  - Research Site, Ústí nad Labem
  - Research Site, Ústí nad Orlicí
  - Research Site, Zábřeh nad Odrou
  - Research Site, Znojmo
- France (23):
  - Research Site, Abbeville
  - Research Site, Albi
  - Research Site, Angers
  - Research Site, Avignon
  - Research Site, Bayonne
  - Research Site, Cannes
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, Jossigny
  - Research Site, La Rochelle
  - Research Site, Le Chesnay
  - Research Site, Le Coudray
  - Research Site, Limoges
  - Research Site, Marseille
  - Research Site, Metz
  - Research Site, Nice
  - Research Site, Nîmes
  - Research Site, Orléans
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Poitiers
  - Research Site, Toulouse
  - Research Site, Tourcoing
- Germany (25):
  - Research Site, Bad Krozingen
  - Research Site, Bad Mergentheim
  - Research Site, Bad Nauheim
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Coburg
  - Research Site, Deggingen
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Esslingen am Neckar
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Kassel
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, Limburg
  - Research Site, Ludwigshafen
  - Research Site, Lübeck
  - Research Site, Mainz
  - Research Site, Mönchengladbach
  - Research Site, Ulm
  - Research Site, Warendorf
  - Research Site, Witten
- Hungary (18):
  - Research Site, Ballasagyarmat
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Debrecen
  - Research Site, Eger
  - Research Site, Gyula
  - Research Site, Kalocsa
  - Research Site, Kecskemét
  - Research Site, Mosonmagyaróvár
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Sopron
  - Research Site, Szeged
  - Research Site, Szekszárd
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
  - Research Site, Zalaegerszeg
- Italy (28):
  - Research Site, Albano Laziale
  - Research Site, Bari
  - Research Site, Benevento
  - Research Site, Brescia
  - Research Site, Carpi
  - Research Site, Catania
  - Research Site, Genova
  - Research Site, Legnano
  - Research Site, Lucca
  - Research Site, Massa
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Osio Sotto Frazione Di Zingoni
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Perugia
  - Research Site, Pescara
  - Research Site, Pisa
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, S Maria Capua Vetere
  - Research Site, Sanremo
  - Research Site, Sassari
  - Research Site, Sessa Aurunca
  - Research Site, Siena
  - Research Site, Sorrento NA
  - Research Site, Vimercate
- Japan (50):
  - Research Site, Akishima-shi
  - Research Site, Amagasaki-shi
  - Research Site, Beppu-shi
  - Research Site, Chūōku
  - Research Site, Daito-shi
  - Research Site, Fukui-shi
  - Research Site, Funabashi-shi
  - Research Site, Gifu
  - Research Site, Hamamatsu
  - Research Site, Himeji-shi
  - Research Site, Imabari
  - Research Site, Isehara-shi
  - Research Site, Kamogawa-shi
  - Research Site, Kanazawa
  - Research Site, Kawachinagano-shi
  - Research Site, Kisarazu-shi
  - Research Site, Komatsushima-shi
  - Research Site, Koriyama-shi
  - Research Site, Kumamoto
  - Research Site, Kure-shi
  - Research Site, Kusatsu-shi
  - Research Site, Kyoto
  - Research Site, Maebashi
  - Research Site, Matsue
  - Research Site, Matsumoto-shi
  - Research Site, Matsuyama
  - Research Site, Meguro-ku
  - Research Site, Miyazaki
  - Research Site, Osaka
  - Research Site, Saga
  - Research Site, Sagamihara-shi
  - Research Site, Saitama-shi
  - Research Site, Sakaide-shi
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Sayama-shi
  - Research Site, Shimada-shi
  - Research Site, Shinagawa-ku
  - Research Site, Shizuoka
  - Research Site, Suwa-shi
  - Research Site, Takarazuka-shi
  - Research Site, Takasaki-shi
  - Research Site, Takatsuki-shi
  - Research Site, Tomakomai-shi
  - Research Site, Toyonaka-shi
  - Research Site, Ueda-shi
  - Research Site, Wakayama
  - Research Site, Wako-shi
  - Research Site, Yatsushiro-shi
  - Research Site, Yokohama
- Netherlands (36):
  - Research Site, Almere Stad
  - Research Site, Amersfoort
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Beverwijk
  - Research Site, Breda
  - Research Site, Delft
  - Research Site, Den Helder
  - Research Site, Deventer
  - Research Site, Drachten
  - Research Site, Ede
  - Research Site, Eindhoven
  - Research Site, Goes
  - Research Site, Groningen
  - Research Site, Hardenberg
  - Research Site, Heerenveen
  - Research Site, Heerlen
  - Research Site, Helmond
  - Research Site, Hilversum
  - Research Site, Hoofddorp
  - Research Site, Hoogeveen
  - Research Site, Leiderdorp
  - Research Site, Maastricht
  - Research Site, Nieuwegein
  - Research Site, Nijmegen
  - Research Site, Oss
  - Research Site, Roosendaal
  - Research Site, Rotterdam
  - Research Site, Schiedam
  - Research Site, Shertogenbosch
  - Research Site, Sittardgeleen
  - Research Site, Sneek
  - Research Site, The Hague
  - Research Site, Tiel
  - Research Site, Tilburg
  - Research Site, Veldhoven
- Norway (11):
  - Research Site, Bergen
  - Research Site, Bodø
  - Research Site, Flekkefjord
  - Research Site, Hamar
  - Research Site, Levanger
  - Research Site, Lillehammer
  - Research Site, Nesttun
  - Research Site, Oslo
  - Research Site, Skien
  - Research Site, Tromsø
  - Research Site, Tynset
- Peru (5):
  - Research Site, Arequipa
  - Research Site, Callao
  - Research Site, Lima
  - Research Site, San Borja
  - Research Site, Trujillo
- Philippines (11):
  - Research Site, Cebu City
  - Research Site, Fuente Osmena Cebu City
  - Research Site, Iloilo City
  - Research Site, Las Piñas
  - Research Site, Lipa City
  - Research Site, Mandaluyong
  - Research Site, Manila
  - Research Site, Pasig
  - Research Site, Quezon
  - Research Site, Quezon City
  - Research Site, San Juan City
- Poland (30):
  - Research Site, Bialystok
  - Research Site, Bielsko-Biala
  - Research Site, Bydgoszcz
  - Research Site, Chorzów
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Giżycko
  - Research Site, Krakow
  - Research Site, Legnica
  - Research Site, Lodz
  - Research Site, Lubin
  - Research Site, Nowa Sól
  - Research Site, Olsztyn
  - Research Site, Opole
  - Research Site, Ostrów Mazowiecka
  - Research Site, Oława
  - Research Site, Piotrków
  - Research Site, Poznan
  - Research Site, Płock
  - Research Site, Skierniewice
  - Research Site, Sobótka
  - Research Site, Sokółka
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Włocławek
  - Research Site, Łańcut
  - Research Site, Łęczna
- Romania (15):
  - Research Site, Bacau
  - Research Site, Brasov
  - Research Site, Brăila
  - Research Site, Bucharest
  - Research Site, Buzău
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Deva
  - Research Site, Focşani
  - Research Site, Iași
  - Research Site, Piteşti
  - Research Site, Sibiu
  - Research Site, Suceava
  - Research Site, Tg. Mures
  - Research Site, Timișoara
- Russia (13):
  - Research Site, Gatchina
  - Research Site, Kazan'
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Perm
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, StPetersburg
  - Research Site, Vladikavkaz
  - Research Site, Volgograd
  - Research Site, Yekaterinburg
- Slovakia (16):
  - Research Site, Banská Bystrica
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Komárno
  - Research Site, Košice
  - Research Site, Liptovský Hrádok
  - Research Site, Liptovský Mikuláš
  - Research Site, Martin
  - Research Site, Nitra
  - Research Site, Partizánske
  - Research Site, Piešťany
  - Research Site, Považská Bystrica
  - Research Site, Prešov
  - Research Site, Ružomberok
  - Research Site, Trnava
  - Research Site, Žilina
- South Africa (15):
  - Research Site, Alberton
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Centurion
  - Research Site, Durban
  - Research Site, Gatesville
  - Research Site, George
  - Research Site, Johannesburg
  - Research Site, Kempron Park
  - Research Site, Panorama
  - Research Site, Parow
  - Research Site, Pretoria
  - Research Site, Somerset West
  - Research Site, Soweto
  - Research Site, Worcester
- South Korea (12):
  - Research Site, Bucheon-si
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gwangju
  - Research Site, Jeonju
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Uijeongbu-si
  - Research Site, Wŏnju
- Spain (16):
  - Research Site, Almería
  - Research Site, Avilés
  - Research Site, Barcelona
  - Research Site, Bilbao
  - Research Site, Don Benito (Badajoz)
  - Research Site, Hospitalet de Llobregat(Barcel
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Oviedo
  - Research Site, Palma de Mallorca
  - Research Site, Sabadell
  - Research Site, San Sebastián de los Reyes
  - Research Site, Santiago(A Coruña)
  - Research Site, Seville
  - Research Site, Valencia
- Sweden (13):
  - Research Site, Eksjö
  - Research Site, Gothenburg
  - Research Site, Jönköping
  - Research Site, Linköping
  - Research Site, Ljungby
  - Research Site, Lund
  - Research Site, Mölndal
  - Research Site, Örebro
  - Research Site, Östersund
  - Research Site, Stockholm
  - Research Site, Sundsvall
  - Research Site, Umeå
  - Research Site, Västerås
- Turkey (Türkiye) (6):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Malatya
  - Research Site, Mersin
- Ukraine (9):
  - Research Site, Dnipro
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Uzhhorod
  - Research Site, Vinnitsa
  - Research Site, Zaporozye
- United Kingdom (23):
  - Research Site, Airdrie
  - Research Site, Antrim
  - Research Site, Belfast
  - Research Site, Blackpool
  - Research Site, Bournemouth
  - Research Site, Brighton
  - Research Site, Bristol
  - Research Site, Coventry
  - Research Site, Dundee
  - Research Site, East Kilbride
  - Research Site, Ely
  - Research Site, Hastings
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Middlesbrough
  - Research Site, Northampton
  - Research Site, Nottingham
  - Research Site, Peterborough
  - Research Site, Rotherham
  - Research Site, Sheffield
  - Research Site, Swansea
  - Research Site, Torquay
  - Research Site, York

REFERENCES:
- [Result] Bonaca MP, Bhatt DL, Cohen M, Steg PG, Storey RF, Jensen EC, Magnani G, Bansilal S, Fish MP, Im K, Bengtsson O, Oude Ophuis T, Budaj A, Theroux P, Ruda M, Hamm C, Goto S, Spinar J, Nicolau JC, Kiss RG, Murphy SA, Wiviott SD, Held P, Braunwald E, Sabatine MS; PEGASUS-TIMI 54 Steering Committee and Investigators. Long-term use of ticagrelor in patients with prior myocardial infarction. N Engl J Med. 2015 May 7;372(19):1791-800. doi: 10.1056/NEJMoa1500857. Epub 2015 Mar 14. PMID 25773268
- [Derived] Bonaca MP, Im K, Magnani G, Bansilal S, Dellborg M, Storey RF, Bhatt DL, Steg PG, Cohen M, Johanson P, Braunwald E, Sabatine MS. Patient selection for long-term secondary prevention with ticagrelor: insights from PEGASUS-TIMI 54. Eur Heart J. 2022 Dec 21;43(48):5037-5044. doi: 10.1093/eurheartj/ehac402. PMID 36367709
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Bergmark BA, Bhatt DL, Steg PG, Budaj A, Storey RF, Gurmu Y, Kuder JF, Im K, Magnani G, Oude Ophuis T, Hamm C, Spinar J, Kiss RG, Van de Werf FJ, Montalescot G, Johanson P, Braunwald E, Sabatine MS, Bonaca MP. Long-Term Ticagrelor in Patients With Prior Coronary Stenting in the PEGASUS-TIMI 54 Trial. J Am Heart Assoc. 2021 Sep 7;10(17):e020446. doi: 10.1161/JAHA.120.020446. Epub 2021 Aug 21. PMID 34423649
- [Derived] Magnani G, Ardissino D, Im K, Budaj A, Storey RF, Steg PG, Bhatt DL, Cohen M, Oude Ophius T, Goudev A, Parkhomenko A, Kamensky G, Angiolillo DJ, Lopez-Sendon J, Johanson P, Braunwald E, Sabatine MS, Bonaca MP. Predictors, Type, and Impact of Bleeding on the Net Clinical Benefit of Long-Term Ticagrelor in Stable Patients With Prior Myocardial Infarction. J Am Heart Assoc. 2021 Feb 16;10(4):e017008. doi: 10.1161/JAHA.120.017008. Epub 2021 Feb 9. PMID 33559485
- [Derived] Furtado RHM, Venkateswaran RV, Nicolau JC, Gurmu Y, Bhatt DL, Storey RF, Steg PG, Magnani G, Goto S, Dellborg M, Kamensky G, Isaza D, Aylward P, Johanson P, Bonaca MP. Caffeinated Beverage Intake, Dyspnea With Ticagrelor, and Cardiovascular Outcomes: Insights From the PEGASUS-TIMI 54 Trial. J Am Heart Assoc. 2020 May 18;9(10):e015785. doi: 10.1161/JAHA.119.015785. Epub 2020 May 15. PMID 32410485
- [Derived] Gencer B, Li XS, Gurmu Y, Bonaca MP, Morrow DA, Cohen M, Bhatt DL, Steg PG, Storey RF, Johanson P, Wang Z, Hazen SL, Sabatine MS. Gut Microbiota-Dependent Trimethylamine N-oxide and Cardiovascular Outcomes in Patients With Prior Myocardial Infarction: A Nested Case Control Study From the PEGASUS-TIMI 54 Trial. J Am Heart Assoc. 2020 May 18;9(10):e015331. doi: 10.1161/JAHA.119.015331. Epub 2020 May 5. PMID 32366163
- [Derived] Furtado RHM, Nicolau JC, Magnani G, Im K, Bhatt DL, Storey RF, Steg PG, Spinar J, Budaj A, Kontny F, Corbalan R, Kiss RG, Abola MT, Johanson P, Jensen EC, Braunwald E, Sabatine MS, Bonaca MP. Long-term ticagrelor for secondary prevention in patients with prior myocardial infarction and no history of coronary stenting: insights from PEGASUS-TIMI 54. Eur Heart J. 2020 May 1;41(17):1625-1632. doi: 10.1093/eurheartj/ehz821. PMID 31811715
- [Derived] Dellborg M, Bonaca MP, Storey RF, Steg PG, Im KA, Cohen M, Bhatt DL, Oude Ophuis T, Budaj A, Hamm C, Spinar J, Kiss RG, Lopez-Sendon J, Kamensky G, Van de Werf F, Ardissino D, Kontny F, Montalescot G, Johanson P, Bengtsson O, Himmelmann A, Braunwald E, Sabatine MS. Efficacy and safety with ticagrelor in patients with prior myocardial infarction in the approved European label: insights from PEGASUS-TIMI 54. Eur Heart J Cardiovasc Pharmacother. 2019 Oct 1;5(4):200-206. doi: 10.1093/ehjcvp/pvz020. PMID 31218354
- [Derived] Bonaca MP, Wiviott SD, Morrow DA, Steg PG, Hamm C, Bhatt DL, Storey RF, Cohen M, Kuder J, Im K, Magnani G, Budaj A, Nicolau JC, Parkhomenko A, Lopez-Sendon J, Dellborg M, Diaz R, Van de Werf F, Corbalan R, Goudev A, Jensen EC, Johanson P, Braunwald E, Sabatine MS. Reduction in Subtypes and Sizes of Myocardial Infarction With Ticagrelor in PEGASUS-TIMI 54. J Am Heart Assoc. 2018 Nov 20;7(22):e009260. doi: 10.1161/JAHA.118.009260. PMID 30571502
- [Derived] Bansilal S, Bonaca MP, Cornel JH, Storey RF, Bhatt DL, Steg PG, Im K, Murphy SA, Angiolillo DJ, Kiss RG, Parkhomenko AN, Lopez-Sendon J, Isaza D, Goudev A, Kontny F, Held P, Jensen EC, Braunwald E, Sabatine MS, Oude Ophuis AJ. Ticagrelor for Secondary Prevention of Atherothrombotic Events in Patients With Multivessel Coronary Disease. J Am Coll Cardiol. 2018 Feb 6;71(5):489-496. doi: 10.1016/j.jacc.2017.11.050. PMID 29406853
- [Derived] Cavallari I, Morrow DA, Creager MA, Olin J, Bhatt DL, Steg PG, Storey RF, Cohen M, Scirica BS, Piazza G, Goodrich EL, Braunwald E, Sabatine MS, Bonaca MP. Frequency, Predictors, and Impact of Combined Antiplatelet Therapy on Venous Thromboembolism in Patients With Symptomatic Atherosclerosis. Circulation. 2018 Feb 13;137(7):684-692. doi: 10.1161/CIRCULATIONAHA.117.031062. Epub 2017 Oct 30. PMID 29084737
- [Derived] Bonaca MP, Storey RF, Theroux P, Steg PG, Bhatt DL, Cohen MC, Im K, Murphy SA, Magnani G, Ophuis TO, Rudah M, Parkhomenko A, Isaza D, Kamensky G, Goudev A, Montalescot G, Jensen EC, Johanson P, Braunwald E, Sabatine MS. Efficacy and Safety of Ticagrelor Over Time in Patients With Prior MI in PEGASUS-TIMI 54. J Am Coll Cardiol. 2017 Sep 12;70(11):1368-1375. doi: 10.1016/j.jacc.2017.07.768. PMID 28882235
- [Derived] Magnuson EA, Li H, Wang K, Vilain K, Shafiq A, Bonaca MP, Bhatt DL, Cohen M, Steg PG, Storey RF, Braunwald E, Sabatine MS, Cohen DJ; PEGASUS-TIMI 54 Trial Investigators. Cost-Effectiveness of Long-Term Ticagrelor in Patients With Prior Myocardial Infarction: Results From the PEGASUS-TIMI 54 Trial. J Am Coll Cardiol. 2017 Aug 1;70(5):527-538. doi: 10.1016/j.jacc.2017.05.063. PMID 28750695
- [Derived] Thomas MR, Angiolillo DJ, Bonaca MP, Ajjan RA, Judge HM, Rollini F, Franchi F, Ahsan AJ, Bhatt DL, Kuder JF, Steg PG, Cohen M, Muthusamy R, Sabatine MS, Storey RF. Consistent platelet inhibition with ticagrelor 60 mg twice-daily following myocardial infarction regardless of diabetes status. Thromb Haemost. 2017 May 3;117(5):940-947. doi: 10.1160/TH16-09-0703. Epub 2017 Mar 16. PMID 28300867
- [Derived] Bonaca MP, Goto S, Bhatt DL, Steg PG, Storey RF, Cohen M, Goodrich E, Mauri L, Ophuis TO, Ruda M, Spinar J, Seung KB, Hu D, Dalby AJ, Jensen E, Held P, Morrow DA, Braunwald E, Sabatine MS. Prevention of Stroke with Ticagrelor in Patients with Prior Myocardial Infarction: Insights from PEGASUS-TIMI 54 (Prevention of Cardiovascular Events in Patients With Prior Heart Attack Using Ticagrelor Compared to Placebo on a Background of Aspirin-Thrombolysis in Myocardial Infarction 54). Circulation. 2016 Sep 20;134(12):861-71. doi: 10.1161/CIRCULATIONAHA.116.024637. Epub 2016 Aug 30. PMID 27576775
- [Derived] Bonaca MP, Bhatt DL, Oude Ophuis T, Steg PG, Storey R, Cohen M, Kuder J, Im K, Magnani G, Budaj A, Theroux P, Hamm C, Spinar J, Kiss RG, Dalby AJ, Medina FA, Kontny F, Aylward PE, Jensen EC, Held P, Braunwald E, Sabatine MS. Long-term Tolerability of Ticagrelor for the Secondary Prevention of Major Adverse Cardiovascular Events: A Secondary Analysis of the PEGASUS-TIMI 54 Trial. JAMA Cardiol. 2016 Jul 1;1(4):425-32. doi: 10.1001/jamacardio.2016.1017. PMID 27438319
- [Derived] Held P, Himmelmann A, Ditmarsch M. Ticagrelor for the treatment of atherosclerotic disease: insights from the PARTHENON clinical development program. Future Cardiol. 2016 Jul;12(4):405-18. doi: 10.2217/fca-2016-0028. Epub 2016 May 10. PMID 27160944
- [Derived] Bonaca MP, Bhatt DL, Storey RF, Steg PG, Cohen M, Kuder J, Goodrich E, Nicolau JC, Parkhomenko A, Lopez-Sendon J, Dellborg M, Dalby A, Spinar J, Aylward P, Corbalan R, Abola MTB, Jensen EC, Held P, Braunwald E, Sabatine MS. Ticagrelor for Prevention of Ischemic Events After Myocardial Infarction in Patients With Peripheral Artery Disease. J Am Coll Cardiol. 2016 Jun 14;67(23):2719-2728. doi: 10.1016/j.jacc.2016.03.524. Epub 2016 Apr 1. PMID 27046162
- [Derived] Bhatt DL, Bonaca MP, Bansilal S, Angiolillo DJ, Cohen M, Storey RF, Im K, Murphy SA, Held P, Braunwald E, Sabatine MS, Steg PG. Reduction in Ischemic Events With Ticagrelor in Diabetic Patients With Prior Myocardial Infarction in PEGASUS-TIMI 54. J Am Coll Cardiol. 2016 Jun 14;67(23):2732-2740. doi: 10.1016/j.jacc.2016.03.529. Epub 2016 Apr 1. PMID 27046160
- [Derived] Bonaca MP, Bhatt DL, Steg PG, Storey RF, Cohen M, Im K, Oude Ophuis T, Budaj A, Goto S, Lopez-Sendon J, Diaz R, Dalby A, Van de Werf F, Ardissino D, Montalescot G, Aylward P, Magnani G, Jensen EC, Held P, Braunwald E, Sabatine MS. Ischaemic risk and efficacy of ticagrelor in relation to time from P2Y12 inhibitor withdrawal in patients with prior myocardial infarction: insights from PEGASUS-TIMI 54. Eur Heart J. 2016 Apr 7;37(14):1133-42. doi: 10.1093/eurheartj/ehv531. Epub 2015 Oct 21. PMID 26491109
- [Derived] Bonaca MP, Bhatt DL, Braunwald E, Cohen M, Steg PG, Storey RF, Held P, Jensen EC, Sabatine MS. Design and rationale for the Prevention of Cardiovascular Events in Patients With Prior Heart Attack Using Ticagrelor Compared to Placebo on a Background of Aspirin-Thrombolysis in Myocardial Infarction 54 (PEGASUS-TIMI 54) trial. Am Heart J. 2014 Apr;167(4):437-444.e5. doi: 10.1016/j.ahj.2013.12.020. Epub 2014 Jan 6. PMID 24655690
- See also: D5132C00001_Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=489&filename=D5132C00001_CSP1.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Participant Flow shows patients randomized. This number is different from patients enrolled in the protocol section which includes patients who were enrolled, but not randomized.
Groups:
- Ticagrelor 90 mg: Ticagrelor 90 mg twice daily (BD)
- Ticagrelor 60 mg: Ticagrelor 60 mg twice daily (BD)
- Placebo: Matching placebo
Period: Overall Study
Arm/Group | Ticagrelor 90 mg | Ticagrelor 60 mg | Placebo
Started | 7050 | 7045 | 7067
Completed | 6995 | 6989 | 7014
Not Completed | 55 | 56 | 53
Not completed — Withdrawal by Subject | 52 | 50 | 52
Not completed — Lost to Follow-up | 3 | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor 90 mg | Ticagrelor 60 mg | Placebo | Total
Number analyzed (Participants) | 7050 | 7045 | 7067 | 21162
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (8.4) | 65.2 (8.4) | 65.4 (8.3) | 65.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1682 | 1661 | 1717 | 5060
  Male | 5368 | 5384 | 5350 | 16102

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of the Percentage of Patients Who Experienced Cardiovascular Death (CV Death), Myocardial Infarction (MI) or Stroke Within 3 Years From Randomization
Description: Participants with CV death, MI or Stroke. If no event, censoring occurs at the earliest of the efficacy cut-off date 14 Sep 2014, withdrawal of consent, non-CV death or at the last time point of complete clinical event assessment. Events were adjudicated by a blinded endpoint committee. The Kaplan-Meier estimate reports the percentage of patients who experienced CV Death, MI or stroke within 3 years from randomization
Time Frame: Randomization up to 47 months
Population: Intention to treat (ITT) population defined as all participants who were randomized to study treatment
Measure: Number; unit: Percentage of Patients
Arm/Group | Ticagrelor 90 mg | Ticagrelor 60 mg | Placebo
Number analyzed (Participants) | 7050 | 7045 | 7067
Percentage of Patients | 7.8 | 7.8 | 9.0
Statistical Analysis 1: Comparison: Ticagrelor 90 mg vs Placebo; Test type: Superiority or Other; p = 0.0080, Regression, Cox; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.75 to 0.96] — The hazard ratio shows ticagrelor 90 mg hazard / placebo hazard
Statistical Analysis 2: Comparison: Ticagrelor 60 mg vs Placebo; Test type: Superiority or Other; p = 0.0043, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.74 to 0.95] — The hazard ratio shows ticagrelor 60 mg hazard / placebo hazard

2. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Patients Who Experienced Cardiovascular Death (CV Death) Within 3 Years From Randomization
Description: Participants with CV death. If no event, censoring occurs at the earliest of the efficacy cut-off date 14 Sep 2014, withdrawal of consent, non-CV death or at the last time point of complete clinical event assessment. Events were adjudicated by a blinded endpoint committee. The Kaplan-Meier estimate reports the percentage of patients who experienced CV Death within 3 years from randomization
Time Frame: Randomization up to 47 months
Population: Intention to treat (ITT) population defined as all participants who were randomized to study treatment
Measure: Number; unit: Percentage of Patients
Arm/Group | Ticagrelor 90 mg | Ticagrelor 60 mg | Placebo
Number analyzed (Participants) | 7050 | 7045 | 7067
Percentage of Patients | 2.9 | 2.9 | 3.4
Statistical Analysis 1: Comparison: Ticagrelor 90 mg vs Placebo; Test type: Superiority or Other; p = 0.1547, Regression, Cox; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.71 to 1.06] — The hazard ratio shows ticagrelor 90 mg hazard / placebo hazard
Statistical Analysis 2: Comparison: Ticagrelor 60 mg vs Placebo; Test type: Superiority or Other; p = 0.0676, Regression, Cox; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.68 to 1.01] — The hazard ratio shows ticagrelor 60 mg hazard / placebo hazard

3. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Patients Who Died From Any Cause Within 3 Years From Randomization
Description: Participants with death from any cause. If no event, censoring occurs at the earliest of the efficacy cut-off date 14 Sep 2014, withdrawal of consent or the last time point the particapant was known to be alive. Events were adjudicated by a blinded endpoint committee. The Kaplan-Meier estimate reports the percentage of patients who died from any cause within 3 years from randomization
Time Frame: Randomization up to 47 months
Population: Intention to treat (ITT) population defined as all participants who were randomized to study treatment
Measure: Number; unit: Percentage of Patients
Arm/Group | Ticagrelor 90 mg | Ticagrelor 60 mg | Placebo
Number analyzed (Participants) | 7050 | 7045 | 7067
Percentage of Patients | 5.1 | 4.7 | 5.2
Statistical Analysis 1: Comparison: Ticagrelor 90 mg vs Placebo; Test type: Superiority or Other; p = 0.9851, Regression, Cox; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.86 to 1.16] — The hazard ratio shows ticagrelor 90 mg hazard / placebo hazard
Statistical Analysis 2: Comparison: Ticagrelor 60 mg vs Placebo; Test type: Superiority or Other; p = 0.1350, Regression, Cox; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.76 to 1.04] — The hazard ratio shows ticagrelor 60 mg hazard / placebo hazard

4. Primary Outcome: Kaplan-Meier Estimate of the Percentage of Patients Who Experienced a TIMI Major Bleeding Within 3 Years From First Dose of Study Drug Units: Percentage of Patients
Description: A Thrombolysis in Myocardial Infarction (TIMI) study group major bleeding is defined as any fatal bleeding (leading directly to death within 7 days), any intrcranial bleeding or any clinically overt signs of haemorrhage associated with a drop in Haemoglobin of >= 5g/dL. Events were adjudicated by a clinical events committee. Censoring ocurrs at 7 days following last dose of study drug. The Kaplan-Meier estimate reports the percentage of patients who experienced a TIMI Major bleeding within 3 years from first dose of study drug
Time Frame: First dosing up to 48 months
Population: The safety analysis set defined as all patients who took at least one dose of study drug
Measure: Number; unit: Percentage of Patients
Arm/Group | Ticagrelor 90 mg | Ticagrelor 60 mg | Placebo
Number analyzed (Participants) | 6988 | 6958 | 6996
Percentage of Patients | 2.6 | 2.3 | 1.1
Statistical Analysis 1: Comparison: Ticagrelor 90 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 2.69, 95% CI 2-sided [1.96 to 3.70] — The hazard ratio shows ticagrelor 90 mg hazard / placebo hazard
Statistical Analysis 2: Comparison: Ticagrelor 60 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 2.32, 95% CI 2-sided [1.68 to 3.21] — The hazard ratio shows ticagrelor 60 mg hazard / placebo hazard

ADVERSE EVENTS:
Description: Adverse events are reported for the safety analysis set, that is patients who received at least one dose of study drug. Hence the number of participants at risk is different from the total number in Participant Flow, which includes all randomized patients.
Arm/Group | Placebo | Ticagrelor 60mg bd | Ticagrelor 90mg bd
Serious Adverse Events (participants affected / at risk) | 1757/6996 | 1853/6958 | 1918/6988
Other Adverse Events (participants affected / at risk) | 945/6996 | 1992/6958 | 2245/6988
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6996) | Ticagrelor 60mg bd (N=6958) | Ticagrelor 90mg bd (N=6988)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 5 (5) | 12 (12)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (7)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Aplastic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Coagulation factor deficiency (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 (2) | 7 (7) | 4 (4)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (3) | 11 (11) | 24 (25)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (5) | 4 (4)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 2 (2)
Pernicious anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Spontaneous haematoma (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 2 (2)
Spontaneous haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 2 (2) | 8 (8)
Acute coronary syndrome (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 5 (6) | 1 (1) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 28 (28) | 20 (20) | 19 (19)
Adams-Stokes syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 51 (53) | 45 (47) | 51 (55)
Angina unstable (Cardiac disorders) | 3 (3) | 2 (2) | 4 (4)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 2 (3) | 3 (3)
Arrhythmia (Cardiac disorders) | 1 (1) | 3 (3) | 2 (2)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 67 (73) | 94 (104) | 74 (88)
Atrial flutter (Cardiac disorders) | 16 (20) | 14 (15) | 13 (13)
Atrial tachycardia (Cardiac disorders) | 4 (4) | 2 (2) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 5 (5) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 13 (14) | 6 (6) | 3 (3)
Atrioventricular block second degree (Cardiac disorders) | 5 (5) | 3 (3) | 4 (4)
Bifascicular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Bradycardia (Cardiac disorders) | 2 (2) | 7 (7) | 7 (7)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 6 (6) | 8 (8) | 7 (8)
Cardiac asthma (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 58 (73) | 53 (70) | 54 (69)
Cardiac failure acute (Cardiac disorders) | 6 (6) | 6 (6) | 4 (4)
Cardiac failure chronic (Cardiac disorders) | 14 (16) | 11 (19) | 19 (25)
Cardiac failure congestive (Cardiac disorders) | 51 (60) | 53 (79) | 70 (97)
Cardiac hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac perforation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 7 (7) | 6 (6) | 6 (7)
Cardiogenic shock (Cardiac disorders) | 10 (10) | 9 (9) | 4 (5)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cor pulmonale chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 6 (6) | 8 (8) | 6 (6)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 3 (3) | 2 (2) | 6 (6)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Dressler's syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Gastrocardiac syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Heart valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (2) | 1 (1) | 8 (8)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Left ventricular failure (Cardiac disorders) | 4 (4) | 1 (1) | 4 (4)
Low cardiac output syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Mitral valve calcification (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 4 (4) | 7 (8) | 0 (0)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial fibrosis (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 11 (11) | 9 (9) | 10 (10)
Myocardial ischaemia (Cardiac disorders) | 3 (3) | 1 (1) | 3 (4)
Myocardial oedema (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial rupture (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 2 (2) | 1 (2) | 0 (0)
Nodal rhythm (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 3 (3) | 3 (3) | 2 (2)
Pericardial effusion (Cardiac disorders) | 4 (4) | 2 (2) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 1 (1) | 3 (4)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 7 (8) | 7 (7) | 8 (9)
Sinoatrial block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 7 (7) | 7 (7) | 12 (12)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Subendocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 5 (5) | 4 (4) | 4 (4)
Systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 3 (4)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 5 (5) | 0 (0) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 3 (3) | 2 (3) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 4 (4) | 4 (6) | 3 (3)
Ventricular fibrillation (Cardiac disorders) | 9 (9) | 11 (11) | 4 (4)
Ventricular tachycardia (Cardiac disorders) | 12 (12) | 17 (20) | 17 (20)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Auricular perichondritis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Inner ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Presbyacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 7 (8) | 3 (3) | 4 (5)
Vertigo labyrinthine (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 3 (3) | 5 (5) | 6 (7)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 2 (2) | 0 (0) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Toxic nodular goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Blindness unilateral (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 14 (17) | 16 (18) | 10 (11)
Cataract nuclear (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 3 (3) | 1 (1) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Endocrine ophthalmopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 2 (2) | 1 (1)
Macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Open angle glaucoma (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Opsoclonus myoclonus (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Pterygium (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal artery embolism (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 4 (5) | 1 (1) | 3 (3)
Retinal haemorrhage (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Tolosa-Hunt syndrome (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 2 (2) | 3 (3) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 5 (5)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 5 (6) | 7 (7)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Appendiceal mucocoele (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 4 (4) | 5 (7) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) | 9 (9)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 7 (7)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 4 (5) | 2 (2) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 3 (3) | 8 (9)
Diverticulum intestinal (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 (2) | 12 (15) | 11 (12)
Duodenal stenosis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 4 (4) | 5 (5)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 4 (4) | 7 (7) | 7 (7)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Faecalith (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Femoral hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 4 (4) | 6 (7) | 13 (14)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 7 (7) | 14 (14) | 18 (18)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 10 (11) | 8 (9) | 17 (18)
Gastritis atrophic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3)
Gastritis hypertrophic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastroduodenitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Gastrointestinal erosion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 (9) | 15 (15) | 26 (27)
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 3 (3) | 5 (5) | 2 (2)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5)
Gastrointestinal vascular malformation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 (11) | 6 (7) | 11 (11)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (3)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (4)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 5 (5) | 3 (3)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1)
Ileus (Gastrointestinal disorders) | 4 (4) | 4 (5) | 4 (4)
Ileus paralytic (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (12)
Inguinal hernia (Gastrointestinal disorders) | 21 (22) | 26 (27) | 25 (25)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 3 (3) | 5 (5)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 8 (8) | 5 (5) | 12 (12)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 3 (3) | 4 (4)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Melaena (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Oesophageal achalasia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal rupture (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pancreatic duct obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 7 (7) | 6 (7) | 7 (8)
Pancreatitis acute (Gastrointestinal disorders) | 7 (7) | 10 (10) | 8 (8)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Papilla of Vater stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Parotid gland inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proctitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3) | 5 (5)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 6 (6) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue blistering (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 3 (3) | 8 (8) | 3 (3)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 7 (7) | 7 (7)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Volvulus of small bowel (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Asthenia (General disorders) | 1 (1) | 7 (9) | 2 (2)
Cardiac death (General disorders) | 1 (1) | 1 (1) | 1 (1)
Catheter site haemorrhage (General disorders) | 2 (2) | 0 (0) | 3 (4)
Chest discomfort (General disorders) | 2 (2) | 4 (4) | 2 (2)
Chest pain (General disorders) | 4 (4) | 2 (2) | 6 (6)
Death (General disorders) | 42 (42) | 34 (34) | 42 (42)
Device battery issue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Device breakage (General disorders) | 0 (0) | 0 (0) | 1 (1)
Device defective (General disorders) | 0 (0) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 1 (1) | 0 (0) | 3 (3)
Device lead damage (General disorders) | 0 (0) | 0 (0) | 2 (2)
Device lead issue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Device malfunction (General disorders) | 2 (2) | 0 (0) | 3 (3)
Device material issue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 0 (0) | 1 (1)
Drowning (General disorders) | 1 (1) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Euthanasia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 2 (2) | 0 (0)
Hernia obstructive (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 2 (2) | 1 (1) | 3 (3)
Implant site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 2 (2) | 1 (1)
Medical device complication (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 109 (118) | 113 (124) | 115 (122)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 3 (3)
Stent-graft endoleak (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 33 (33) | 27 (27) | 27 (27)
Sudden death (General disorders) | 9 (9) | 11 (11) | 6 (6)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 8 (10) | 7 (8) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary fistula (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Biloma (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 3 (3) | 2 (2) | 3 (3)
Cholangitis sclerosing (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 5 (5) | 17 (17) | 10 (10)
Cholecystitis acute (Hepatobiliary disorders) | 11 (11) | 11 (13) | 7 (7)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 4 (4) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 31 (31) | 18 (18) | 15 (15)
Cholestasis (Hepatobiliary disorders) | 3 (3) | 1 (1) | 0 (0)
Chronic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 3 (3) | 0 (0) | 1 (1)
Hepatic vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatorenal failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrocholecystis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 2 (2) | 0 (0)
Reaction to food additive (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Abdominal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 4 (4)
Abscess neck (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Acquired immunodeficiency syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Amoebiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Appendicitis (Infections and infestations) | 9 (9) | 8 (8) | 7 (7)
Appendicitis perforated (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Arthritis infective (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Avian influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Bacterial prostatitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bartholin's abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 19 (20) | 10 (14) | 22 (27)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Bronchopneumonia (Infections and infestations) | 8 (8) | 6 (6) | 12 (12)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bursitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 14 (15) | 17 (19) | 12 (13)
Cellulitis laryngeal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis of male external genital organ (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cerebral toxoplasmosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cholangitis suppurative (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Clostridium difficile sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Congo-Crimean haemorrhagic fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 3 (3) | 3 (3)
Dengue fever (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 4 (4) | 4 (5) | 2 (2)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Diabetic foot infection (Infections and infestations) | 3 (4) | 2 (2) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 12 (12) | 8 (8) | 11 (12)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Emphysematous cholecystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Encephalitis brain stem (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 1 (1) | 4 (4)
Epiglottitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 7 (7) | 4 (4) | 4 (5)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 8 (8) | 5 (8) | 5 (5)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 18 (18) | 15 (16) | 18 (18)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 4 (4) | 2 (2) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Groin infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
H1N1 influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatitis A (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex meningoencephalitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 3 (3) | 2 (2) | 2 (2)
Incision site infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infected fistula (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Infectious colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 6 (6) | 3 (4) | 2 (2)
Influenza (Infections and infestations) | 4 (4) | 0 (0) | 2 (2)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Leishmaniasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Listeria sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Lobar pneumonia (Infections and infestations) | 4 (4) | 2 (2) | 3 (3)
Localised infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 6 (7) | 4 (4)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Muscle abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Myringitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Nasal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 5 (5) | 7 (7) | 5 (5)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Otitis media chronic (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pancreatic abscess (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Paraspinal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 3 (3) | 3 (3) | 6 (6)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 76 (83) | 69 (72) | 77 (86)
Pneumonia bacterial (Infections and infestations) | 11 (12) | 15 (15) | 6 (6)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 5 (5) | 1 (1) | 1 (1)
Post procedural pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 2 (2) | 8 (9) | 2 (3)
Proctitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 5 (5) | 5 (5) | 4 (4)
Pyelonephritis acute (Infections and infestations) | 2 (4) | 2 (2) | 3 (4)
Pyopneumothorax (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3) | 4 (4)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Retroperitoneal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 15 (16) | 20 (20) | 17 (18)
Septic necrosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 6 (6) | 7 (7) | 12 (12)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 4 (4)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Streptococcal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Subacute endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Toxoplasmosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tuberculosis (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 6 (6) | 1 (1)
Urethritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary bladder abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 15 (15) | 27 (30) | 28 (30)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 5 (5) | 5 (5) | 19 (19)
Vestibular neuronitis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
Viral diarrhoea (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Wound abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 3 (3) | 5 (5) | 6 (7)
Wound infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Yersinia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 (2) | 2 (3) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1)
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Anastomotic complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 4 (4) | 11 (11) | 5 (5)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arterial restenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bone fissure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2)
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 6 (6) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 4 (4)
Femoral neck fracture (Injury, poisoning and procedural complications) | 7 (7) | 7 (7) | 4 (4)
Femur fracture (Injury, poisoning and procedural complications) | 10 (11) | 11 (11) | 11 (11)
Fibula fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4) | 2 (2)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fractured ischium (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gas poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Haematuria traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (5) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2)
Heat exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 7 (7) | 8 (8) | 5 (5)
Humerus fracture (Injury, poisoning and procedural complications) | 4 (4) | 7 (7) | 5 (5)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 4 (4)
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Inflammation of wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint capsule rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 7 (7) | 5 (6)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 4 (4)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 6 (6) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 5 (5)
Multiple fractures (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 2 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
Pancreatic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (2) | 0 (0)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post gastric surgery syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 7 (7) | 4 (4)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 6 (7) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 10 (11) | 8 (8) | 11 (12)
Post procedural persistent drain fluid (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 5 (5) | 6 (7)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radial nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radiation dysphagia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (5) | 5 (5)
Remnant gastritis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Renal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 8 (8) | 5 (5) | 8 (8)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 5 (5) | 2 (2)
Scapula fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 10 (10) | 2 (2) | 4 (4)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 5 (5)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 4 (5) | 4 (4)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 6 (6)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Traumatic haematoma (Injury, poisoning and procedural complications) | 4 (4) | 10 (10) | 13 (14)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 11 (13) | 17 (19) | 18 (20)
Traumatic spinal cord compression (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 3 (3) | 5 (5) | 2 (2)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Urinary tract injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
VIIIth nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Venous injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 0 (0)
Blood electrolytes decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cardiac stress test abnormal (Investigations) | 0 (0) | 0 (0) | 2 (2)
Clostridium test positive (Investigations) | 0 (0) | 0 (0) | 1 (2)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymph node palpable (Investigations) | 0 (0) | 1 (1) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Scan myocardial perfusion abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 8 (8) | 9 (9) | 11 (13)
Diabetes mellitus (Metabolism and nutrition disorders) | 13 (15) | 15 (15) | 15 (17)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 13 (13) | 12 (13) | 11 (14)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (6) | 6 (6) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 3 (4)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 6 (6)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 9 (9) | 5 (5) | 10 (10)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (10) | 8 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hand deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 14 (15) | 10 (10) | 8 (11)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Jaw disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7) | 5 (5)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle hypertrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 20 (20) | 22 (23) | 16 (17)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 59 (62) | 54 (59) | 54 (57)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Resorption bone increased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3) | 12 (12)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (3) | 9 (9) | 3 (3)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 7 (8)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3) | 3 (3)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1)
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Tendon calcification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acinic cell carcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1) | 2 (2)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5) | 3 (3)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 7 (7) | 7 (7)
Adenolymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ameloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Anaplastic large cell lymphoma T- and null-cell types (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Astrocytoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (9) | 4 (4) | 9 (12)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
Benign neoplasm of ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (12) | 15 (15) | 5 (5)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (5) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 7 (7) | 4 (4)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4) | 3 (3)
Bladder transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) | 0 (0)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Bone sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 4 (4) | 7 (7)
Breast cancer male (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (3) | 4 (4)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Brenner tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) | 2 (2)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (4) | 7 (7)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 14 (14) | 14 (14)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 5 (5) | 7 (9)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1) | 2 (2)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Epithelioid mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Follicle centre lymphoma, follicular grade I, II, III stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 2 (2)
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (9) | 6 (6) | 8 (10)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal stromal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2)
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (2)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (3) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0) | 4 (4)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 3 (4)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 11 (11) | 14 (14)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 10 (10) | 17 (17)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 4 (4)
Lymphoma cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lymphoplasmacytoid lymphoma/immunocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (12) | 7 (7) | 5 (5)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 2 (2)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1) | 1 (1)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1) | 2 (2)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 4 (4)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Metastatic salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Nasal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 2 (2)
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Non-Hodgkin's lymphoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma unspecified histology aggressive (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4) | 5 (6)
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oral cavity cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Ovarian cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancoast's tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (3) | 6 (7)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 4 (5) | 5 (5)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Paranasal sinus neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0)
Penis carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3) | 0 (0)
Peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 2 (2)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1)
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 37 (37) | 29 (29) | 38 (38)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5) | 8 (8)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 2 (2)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 3 (3)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5) | 3 (3)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5) | 4 (4)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2) | 5 (5)
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Salivary gland cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Sarcomatoid mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (5) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 4 (4)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Splenic marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 4 (4)
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tongue cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tonsillar neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 6 (6) | 6 (6)
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Undifferentiated nasopharyngeal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Brain stem syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Carotid artery disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 5 (5) | 7 (7) | 15 (17)
Carotid sinus syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebellar ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1)
Cerebral cyst (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 5 (5) | 5 (5) | 2 (2)
Cerebral infarction (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral microangiopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cervical cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cluster headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Complex regional pain syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1)
Dementia (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Demyelinating polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 6 (6) | 9 (10)
Encephalopathy (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1) | 5 (6)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 10 (10) | 3 (3) | 5 (5)
Haemorrhagic transformation stroke (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 4 (4)
Hypercapnic coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
IIIrd nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 18 (19) | 11 (11) | 11 (11)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Mononeuritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nerve root compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Neuritis cranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Occipital neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic intolerance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral nerve paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 6 (6) | 8 (8) | 3 (3)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Quadriparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 3 (3) | 1 (1) | 3 (4)
Senile dementia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Serotonin syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal claudication (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 28 (30) | 31 (33) | 37 (39)
Temporal lobe epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient global amnesia (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Uraemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
VIth nerve paresis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Vagus nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1)
Vascular parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vertebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (3) | 4 (4) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 2 (2) | 0 (0) | 3 (3)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 8 (11) | 8 (8) | 11 (13)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Major depression (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 3 (3) | 2 (2) | 3 (3)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Psychiatric decompensation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychiatric symptom (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Somatoform disorder cardiovascular (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Bladder diverticulum (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Bladder neck sclerosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 2 (2) | 3 (3) | 2 (2)
Calculus ureteric (Renal and urinary disorders) | 4 (4) | 6 (6) | 5 (5)
Calculus urethral (Renal and urinary disorders) | 1 (1) | 1 (1) | 4 (4)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 3 (3) | 2 (2)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (3) | 8 (11) | 9 (9)
Haemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 4 (4)
Hypertensive nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 8 (12) | 10 (11) | 21 (22)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 3 (3) | 4 (4)
Renal cyst (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1)
Renal cyst ruptured (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 15 (18) | 8 (9) | 6 (6)
Renal failure acute (Renal and urinary disorders) | 28 (34) | 32 (32) | 32 (34)
Renal failure chronic (Renal and urinary disorders) | 6 (6) | 7 (8) | 5 (6)
Renal haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 4 (4) | 4 (4) | 1 (1)
Renal tubular acidosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureteric rupture (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 2 (2) | 1 (1) | 3 (3)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary bladder polyp (Renal and urinary disorders) | 2 (2) | 4 (4) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 4 (4) | 3 (3) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinoma (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acquired hydrocele (Reproductive system and breast disorders) | 4 (5) | 4 (4) | 2 (2)
Acquired phimosis (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 26 (26) | 25 (26) | 20 (20)
Breast fibrosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Calculus prostatic (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (2)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Ovarian necrosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0)
Prostatic mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatism (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 7 (7) | 5 (5) | 5 (5)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2)
Uterine cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 2 (3)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2) | 6 (7)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 6 (6) | 9 (12)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 45 (65) | 39 (62) | 54 (74)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diffuse panbronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 23 (24) | 29 (30)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Epiglottic oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 15 (17) | 20 (21)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 5 (6)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 5 (5)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural adhesion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 6 (7) | 2 (3)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 5 (5) | 5 (5)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 17 (17) | 21 (23)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 5 (5) | 5 (5)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7) | 6 (6)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 3 (3)
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3) | 2 (2)
Cutaneous sarcoidosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 4 (4)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry gangrene (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 2 (2)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Angiodysplasia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 13 (13) | 19 (19) | 19 (20)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 0 (0) | 4 (4)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Aortic dissection rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 8 (8) | 2 (2) | 2 (2)
Aortic thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Aorto-duodenal fistula (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial rupture (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 10 (10) | 4 (5) | 10 (11)
Diabetic vascular disorder (Vascular disorders) | 3 (3) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (2) | 0 (0) | 1 (1)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Femoral artery embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 18 (18) | 15 (15) | 8 (8)
Hypertensive crisis (Vascular disorders) | 12 (14) | 8 (8) | 10 (11)
Hypertensive emergency (Vascular disorders) | 1 (1) | 4 (5) | 0 (0)
Hypotension (Vascular disorders) | 10 (10) | 9 (9) | 10 (10)
Hypothenar hammer syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 5 (5) | 4 (4) | 4 (4)
Leriche syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Malignant hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 4 (4) | 4 (4) | 5 (5)
Penetrating atherosclerotic ulcer (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 15 (18) | 10 (10) | 17 (17)
Peripheral artery aneurysm (Vascular disorders) | 3 (3) | 4 (4) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 17 (22) | 5 (7) | 5 (6)
Peripheral artery thrombosis (Vascular disorders) | 5 (5) | 3 (4) | 4 (4)
Peripheral circulatory failure (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral embolism (Vascular disorders) | 1 (1) | 3 (3) | 1 (2)
Peripheral ischaemia (Vascular disorders) | 9 (13) | 3 (3) | 5 (6)
Peripheral vascular disorder (Vascular disorders) | 8 (8) | 1 (1) | 4 (5)
Poor peripheral circulation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Steal syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Subclavian artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Temporal arteritis (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 5 (6) | 2 (2)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Venous insufficiency (Vascular disorders) | 1 (2) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6996) | Ticagrelor 60mg bd (N=6958) | Ticagrelor 90mg bd (N=6988)
Increased tendency to bruise (Blood and lymphatic system disorders) | 65 (70) | 419 (520) | 464 (575)
Nasopharyngitis (Infections and infestations) | 377 (469) | 364 (486) | 368 (490)
Contusion (Injury, poisoning and procedural complications) | 111 (122) | 353 (471) | 385 (473)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 329 (362) | 876 (1036) | 1091 (1340)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 165 (221) | 420 (623) | 505 (668)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No